CLINICAL TRIAL: NCT04518111
Title: Early Clinical Outcome of Medial Unicompartmental Knee Arthroplasty (UKA) and High Tibial Osteotomy (HTO) for the Treatment of Anteromedial Osteoarthritis (AMOA) in Chinese Population
Brief Title: Oxford UKA and HTO Post-market Clinical Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CSA2019-47K
Record Dates: First submitted 2020-08-11; First posted 2020-08-19 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Knee Osteoarthritis
Keywords: Anteromedial osteoarthritis (AMOA)
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Unicompartmental Knee Arthroplasty (UKA): Patients who underwent primary UKA with Oxford Partial Knee with the Microplasty® instrumentation for AMOA.
- High Tibial Osteotomy (HTO): Patients who underwent Open Wedge HTO for AMOA.

SUMMARY:
The purpose of this study is to compare the performance and safety of medial UKA and HTO in the treatment of AMOA in term of functional outcome, radiographic assessment, range of motion, postoperative complications, revision rate and relevant health economics outcome.

DETAILED DESCRIPTION:
The purpose of this study is to compare the outcomes of medial UKA and HTO in the treatment of AMOA by investigating the performance of these 2 procedures in terms of functional outcome, radiographic assessment, range of motion, postoperative complications, revision rate and relevant health economics outcome, then identify factors associated with better clinical performance. It is aimed to provide evidence-based guidelines for selecting the appropriate procedure in managing AMOA in Chinese population based on the findings of this study.

The secondary endpoints will include:

1. Pain Numerical Rating Scale (NRS)
2. SF-12 Health Survey
3. Radiographic assessment includes pre-op and post-op mechanical femorotibial angle (mFTA), patella height, patellofemoral medial and lateral articular surfaces, and displacement angle of patella
4. Range of motion
5. Adverse event rate and classification (including complication)
6. Operating time
7. Total blood loss (BRECHER formula)
8. Revision rate

Health economic outcomes based on hospital discharge days, recovery time, physiotherapy and complications/ reoperations will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is aged 18 to 85 years old, inclusive;
2. Patients who diagnosed with AMOA of the knee, and have undergone Open Wedge HTO, or primary unilateral partial knee arthroplasty with Oxford Partial Knee with Microplasty® instrumentation in accordance to indications of UKA and the following radiographic assessments in the knee joint:

   * exposed bone on both the femur and tibia in the medial compartment.
   * functionally intact ACL
   * full thickness lateral cartilage (ignore osteophytes)
   * functionally normal MCL: correctable deformity (normal medial opening)
   * acceptable patellofemoral joint: normal, medial facet OA with or without bone loss, lateral facet OA without bone loss.
3. UKA or HTO procedure completed one year prior to study participation;
4. Patient provides written informed consent by signing and dating the Institutional Review Board/Ethics Committee (IRB/EC) approved informed consent form.

Exclusion Criteria:

1. Has undergone UKA but met any of the contraindications included in the product labeling of Oxford Partial Knee system;
2. Has rheumatoid arthritis or other forms of inflammatory joint disease;
3. Uncooperative or with neurologic disorders who are incapable of following directions;
4. Has a diagnosed systemic disease that could affect his/her safety or the study outcome;
5. Anterior cruciate ligament and posterior cruciate ligament injury, collateral ligament instability;
6. Known to be pregnant;
7. Prisoner or known alcohol / drug abuser.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent either primary UKA with Oxford Partial Knee with the Microplasty® instrumentation or Open Wedge HTO for AMOA, and meet the inclusion criteria and do not meet any exclusion criteria will be screened to this study.
Sampling Method: Non-Probability Sample
Enrollment: 370 (Estimated)
Dates: Start 2021-04-24 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Oxford Knee Score | 2 years
  Oxford Knee Score is a patient reported outcome measure questionnaire with a total score range from 0 (severe arthritis) to 48 (satisfactory joint function). The questionnaire contains 12 questions, each with five options scoring from 0 to 4 with 4 being the best outcome for each question.

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) | Pre-op, Post-op 1 month, 3 month, 6 month, 1 year and 2 year
  The Numeric Rating Scale (NRS) is a measure of pain intensity in adults that consists of a numeric version of the visual analog scale numbers between 0 and 10 where 0 indicates "no pain" and 10 indicates "maximum pain". Respondents select a whole one number between 0 and 10, which is best representative of their pain intensity with higher scores indicating greater pain intensity.
SF-12 Health Survey | Pre-op, Post-op 1 month, 3 month, 6 month, 1 year and 2 year
  The Short Form-12 Health Survey (SF-12) measures generic health concepts relevant across age, disease, and treatment groups. It was designed to measure general health status from the patient's point of view and includes 8 concepts commonly represented in health surveys: physical functioning, role functioning physical, bodily pain, general health, vitality, social functioning, role functioning emotional, and mental health. Two summary scores are reported from the SF-12, namely a mental component score (MCS-12) and a physical component score (PCS-12). All subscale scores were transformed to a 0 to 100 scale with the higher score indicating less dysfunction, impairment, or pain.
Mechanical femorotibial angle (mFTA) | Pre-op, Post-op 1 month, 3 month, 6 month, 1 year and 2 year
  Mechanical femorotibial angle is a measurement that assess the mechanical alignment of the lower limb using the long-leg radiograph. It is the lesser angle intersecting the mechanical femoral axis (the line from the center of the femoral head to the knee center) and the mechanical tibial axis (the line from the knee center to the ankle center).
Range of motion | Pre-op, Post-op 1 month, 3 month, 6 month, 1 year and 2 year
  Measurement of flexion and extension degree of the affected joint.
Adverse event rate and classification | Intra-op, post-op 1 year and 2 year
  Summary of adverse events recorded during the study period, including complication and reoperation.

CONTACTS AND LOCATIONS:
Overall Officials: Ye Huang, Principal Investigator — Beijing Chaoyang Emergency Medical Center
Locations (1):
- Beijing Chaoyang Emergency Medical Center, Beijing, China

IPD SHARING:
Plan to Share IPD: No